CLINICAL TRIAL: NCT03450330
Title: A Phase I/II, Open-Label, Multicentre Study to Investigate the Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of AZD4205 as Monotherapy or in Combination With Osimertinib in Patients With EGFR Mutant Advanced Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Assessing an Oral Janus Kinase Inhibitor, AZD4205, in Combination With Osimertinib in Patients Who Have Advanced Non-small Cell Lung Cancer
Acronym: JACKPOT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2017J0001
Record Dates: First submitted 2018-01-25; First posted 2018-03-01 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-11

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- daily dose of AZD4205 (Experimental): daily dose of AZD4205
  Interventions: Drug: AZD4205

INTERVENTIONS:
Drug: AZD4205 — Daily dose of AZD4205, followed by daily dose of AZD4205 and Osimertinib 80 mg. Starting dose of AZD4205 at 75 mg, administered once daily. If tolerated, subsequent cohorts will test increasing doses of AZD4205, and in combination with Osimertinib 80 mg.

SUMMARY:
This study will treat patients with advanced NSCLC who have progressed following prior therapy. This is the first time this drug has ever been tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body and preliminarily assess its anti-cancer activity as monotherapy and in combination with Osimertinib.

DETAILED DESCRIPTION:
A phase I/II, open-label, multicentre study to investigate the safety, tolerability, pharmacokinetics and anti-tumour activity of AZD4205 as monotherapy or in combination with Osimertinib in patients with EGFR mutant advanced stage non-small cell lung cancer (NSCLC). This study includes dose escalation part and dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Obtained written informed consent
2. Patients must have histological or cytological confirmation of activating EGFR mutation positive NSCLC and have failed prior EGFR TKIs treatment.
3. Patients must exhibit Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Adequate bone marrow reserve and organ system functions

Exclusion Criteria:

1. Any unsolved toxicity > CTCAE grade 1 from previous anti-cancer therapy (except alopecia)
2. Active viral or bacterial infections;
3. Active or latent tuberculosis;
4. History of interstitial lung disease (ILD)
5. History of heart failure or QT interval prolongation
6. Immunodeficiency diseases;
7. Active CNS metastases
8. Treatment with an EGFR TKI (e.g., erlotinib or gefitinib) within 8 days or approximately 5 x half-life, whichever is longer, of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of AZD4205 | 21 days after the first dose
  Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | RECIST tumour assessments every 6 weeks from enrollment until study completion, an average of 1 year
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (by investigator assessment) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Peak Plasma Concentration (Cmax) of AZD4205 | 1,8,15 days after first dose
  Peak Plasma Concentration (Cmax) of AZD4205
Area under the plasma concentration versus time curve (AUC) of AZD4205 | 1,8,15 days after first dose
  Area under the plasma concentration versus time curve (AUC) of AZD4205

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Yang, MD, PhD, Study Director — Dizal (Jiangsu) Pharmaceutical Co., Ltd.
Locations (4):
- Australia (4):
  - St George Hospital, Sydney, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Northern Cancer Institute St Leonards, Sydney

IPD SHARING:
Plan to Share IPD: No